CLINICAL TRIAL: NCT06593041
Title: ROLE of PLATELETS in the PATHOPHYSIOLOGY of SYSTEMIC LUPUS
Acronym: PLAQUETTOLUP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8974
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus; Systemic Scleroderma Meeting; ANCA Vasculitis; Inflammatory Myositis; Gougerot-Sjögren Syndrome; Rheumatoid Arthritis
Keywords: PLATELETS; PATHOPHYSIOLOGY; SYSTEMIC LUPUS
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples: For each biological check-up carried out as part of routine care, or in case of flare, an additional 25 mL will be punctured for research purposes, if the patient's condition allows.
  * Tissue samples (skin biopsy, kidney biopsy, synovial biopsy and accessory salivary gland biopsy) + Joint, pleural, alveolar and pericardial fluid samples: Remains will be requalified as research if the remaining quantity allows.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- systemic lupus erythematosus patients

SUMMARY:
Blood platelets, well known for their role in hemostasis, are abnormally activated in patients suffering from systemic lupus erythematosus (SLE), but also from other immunomediated diseases (scleroderma, vasculitis, myositis, Gougerot-Sjögren's and rheumatoid arthritis) in cases of high disease activity. Once activated, platelets express adhesion molecules such as P-selectin on their surface, enabling them to interact physically with immune cells. In a recent work, we identified that activated platelets from lupus patients interact with regulatory T cells and block their regulatory function, thus participating in the deregulated activation of the immune system in SLE. In addition, inhibition of platelet-immune cell interactions by an anti-P-selectin antibody improved LES symptoms in two mouse models.

The aim of this work is to investigate other potential platelet-immune cell interactions in patients with SLE, in comparison with other autoimmune diseases (systemic scleroderma, ANCA vasculitides, inflammatory myositis, Gougerot-Sjögren syndrome and rheumatoid arthritis).

This study could lead to a better understanding of the role of platelets in the pathophysiology of autoimmune diseases, identify new biomarkers of activity, and assess the potential of new therapeutic avenues in these diseases, such as platelet targeting.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age
* Patient affiliated to a health insurance scheme (beneficiary or beneficiary's beneficiary)
* Patient able to understand the aims and risks of research
* Patient having signed and dated an informed consent form
* Patient for whom the diagnosis of at least one of the following pathologies has been confirmed:
* Systemic lupus erythematosus meeting ACR/EULAR 20195 classification criteria.
* Systemic scleroderma meeting ACR/EULAR 20136 classification criteria.
* ANCA vasculitis according to EULAR/ACR 2022.7-9 classification criteria.
* Inflammatory myositis according to EULAR/ACR 201710 classification criteria.
* Gougerot-Sjögren syndrome according to EULAR/ACR 2016 classification criteria11.
* Rheumatoid arthritis according to ACR/EULAR 201012 classification criteria.

Exclusion Criteria:

* Patient in exclusion period (determined by a previous or current study)
* Inability to give patient informed consent (patient in emergency or immediate life-threatening situation)
* Patient under court protection
* Patient under guardianship or curatorship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic auto-immune disease such as :
  * Systemic lupus
  * Anca-associated vasculitis
  * Sjögren's disease
  * Rheumatoid arthritis
  * Systemic sclerosis
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the percentage of circulating aggregates between platelets and immune cells according to disease activity, assessed by flow cytometry. | Every visit for 3 years

SECONDARY OUTCOMES:
Phenotypic impact of platelet/immune cell interaction. | Every visit (each 6 months) for 3 years
  The impact of platelet/immune cell interaction will be assessed using flow cytometry on patient samples. Using a spectral cytometer (Aurora, Cytek) and a multi-color panel (45 colors), we will study the phenotype and degree of activation of different immune subpopulations according to whether or not they interact with platelets. This analysis will be carried out several times during the different visits, and mirrored with the disease activity criteria studied. Activation molecule expression will be analyzed using the same methods as for the main criterion (comparison of the patient with himself/herself using longitudinal samples).

OTHER OUTCOMES:
Transcriptomic impact of platelet/immune cell interaction. | Every visit (each 6 months) for 3 years
  To understand the impact of platelet/immune cell interaction at a finer level, we will sort several immune subpopulations (neutrophils, plasmacytoid dendritic cells, regulatory T lymphocytes) aggregated (CD41+) or not (CD41-) to platelets from patient samples by flow cytometry. Total RNA will be isolated from these subpopulations and sequenced by RNAsequencing to assess the impact of the interaction on the immune cell transcriptome.
  New techniques such as single-cell RNAseq will be used to assess differences between aggregates and non-aggregates.
Measurement of biomarkers of disease activity / predictive of disease flare-ups. | Every visit (each 6 months) for 3 years
  Identifying the mechanisms by which platelets impact immune cells could enable the development of biomarkers of disease activity or prediction of inflammatory flare-ups. These could be molecules of platelet origin (P-selectin, ß-thrombomodulin) or molecules of immune origin produced following interactions with platelets (cytokines, DAMPs). These molecules will be measured using commercial ELISA kits, and analyzed by the same methods as the primary endpoint (comparison of the patient with himself/herself by longitudinal sampling).
Identification of genetic polymorphisms | Every visit (each 6 months) for 3 years
  Identification of genetic polymorphisms (identified by next-generation sequencing) predisposing to platelet activation and targeted sequencing of genes predisposing to platelet activation (FCGR2A,SELP genes) or immune cell activation in inflammatory diseases (SELPG; CD40LG genes).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbourg - Hopital de Hautepierre - Service de rhumatologie, Strasbourg, France, France

IPD SHARING:
Plan to Share IPD: Undecided